CLINICAL TRIAL: NCT01498380
Title: The Bolus Dose of Dexmedetomidine (ED50) That Avoids Hemodynamic Compromise in Children
Acronym: DexMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Carolyne Montgomery, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11-03137
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2014-02

CONDITIONS: Hemodynamic Instability
Keywords: Dexmedetomidine; Precedex; TIVA; Rapid bolus
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexmedetomidine Rapid Bolus (Experimental): All subjects will receive a rapid bolus of dexmedetomidine following induction of anesthesia with propofol and remifentanil and placement of laryngeal mask airway.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The bolus dose of dexmedetomidine given will range from 0.25-2.0 mcg/kg and will be based on the up-and-down method, such that subject 1 will receive 0.5 mcg/kg and if no significant hemodynamic changes occur (heart rate decrease < 20% or blood pressure decrease/increase < 20%) the does will be increased by 0.25 mcg/kg for the subsequent subject. If significant hemodynamic changes occur (HR decrease >/= 20% or SBP/DBP/MAP decrease or increase >/= 20%) the dose will be decreased by 0.25 mcg/kg for the subsequent subject. Each subject will be observed for 10 minutes following the dexmedetomidine bolus.
  Other Names: Precedex

SUMMARY:
Dexmedetomidine is a sedative drug that has many benefits when given to children under anesthesia, such as improved pain relief and reduced agitation following their surgery. It is usually given as an intravenous infusion over 10 minutes, to avoid the changes in heart rate and blood pressure that are occasionally seen when it is administered more quickly. However, this is often infeasible and usually inconvenient. The investigators aim to determine the dose of dexmedetomidine that can be given rapidly (over 5 seconds) without causing significant changes in heart rate and blood pressure. This will be the only study specific intervention.

DETAILED DESCRIPTION:
Purpose This study is being conducted to determine the dose of dexmedetomidine that can be given as a rapid bolus (over 5 seconds) following induction of anesthesia and insertion of a laryngeal mask airway (LMA) without causing significant hemodynamic compromise in healthy children.

Hypothesis We hypothesize that a rapid bolus of dexmedetomidine does not cause significant hemodynamic effects in healthy children.

Justification Dexmedetomidine given in a single peri-operative bolus without subsequent infusion has been shown to be beneficial. It would be arguably more practical to administer the dose as a rapid bolus. The hemodynamic effects of this have not been previously studied in healthy ASA I-II children (aged 5-10 years).

Objectives The objective of this study is to determine the dose of dexmedetomidine that can be given as a rapid bolus in healthy children following induction of total intravenous anesthesia (TIVA) without causing significant hemodynamic compromise.

Research Method This is a prospective, sequential design study using the up-and-down method (UDM) to determine the dose of dexmedetomidine that will prevent hemodynamic compromise following a rapid bolus in healthy children. The only study specific intervention will be a bolus of dexmedetomidine following induction of TIVA and insertion of an LMA.

Pre-operatively Heart rate (HR), non-invasive blood pressure (NIBP), respiratory rate (RR) and oxygen saturation (SpO2) will be obtained in the SDCU. Topical local anesthesia will be applied to potential cannulation sites.

Intra-operatively Following establishment of intravenous access, induction of anesthesia will proceed with lidocaine 1 mg/kg, propofol 4 mg/kg and remifentanil 2 mcg/kg, administered as a bolus over 5 seconds. Bag mask ventilation with 100% oxygen will then be administered whilst SpO2, electrocardiogram (ECG), NIBP and Bispectral Index (BIS) monitoring is attached. Maintenance of anesthesia will be commenced after 30 seconds, with total intravenous anesthesia (TIVA) prepared as a combined infusion of a fixed concentration of propofol 10 mg/ml and remifentanil 5 mcg/ml (PR5) at a dose of propofol 200 mcg/kg/min and remifentanil 0.1 mcg/kg/min, as is the routine practice at BCCH. If further anesthesia is required, rescue doses of PR5 will be administered as propofol 0.5 mg/kg combined with remifentanil 0.25 mcg/kg until a satisfactory level of anesthesia is reached. Any rescue doses given will be documented. After the maintenance infusion is commenced, a NIBP will be recorded. A pre-programmed bolus dose of 10 ml/kg 0.9% saline will simultaneously be delivered (over 10 minutes) when the maintenance TIVA infusion is commenced. Following this, the intravenous fluid infusion will be programmed to run at maintenance rates according to the weight of the child.

One minute after induction, an LMA will be inserted and secured in place (T0). Positive pressure ventilation will be commenced, or the patient allowed to breathe spontaneously, as appropriate. Supplemental oxygen will be administered as needed to maintain SpO2 ≥ 96%. If further anesthesia is required, rescue doses of PR5 will be administered and documented, as above.

One minute after successful LMA insertion (T1), a NIBP recording will be taken, along with a baseline HR that will be being monitored continuously. This will constitute the baseline NIBP and HR (pre-study drug intervention) and will be used to define changes in hemodynamics of systolic, mean, diastolic blood pressure (SBP, MAP and DBP, respectively) and HR following the study drug intervention.

One minute after the baseline NIBP is recorded, a bolus dose of dexmedetomidine will be administered over 5 seconds (T2). The dose will be dictated by the UDM study design, with a starting dose of 0.5 mcg/kg. The dexmedetomidine will be diluted in 0.9% saline to achieve the required concentration of 4 mcg/ml prior to administration. NIBP readings will be recorded every minute following the bolus, for a period of 10 minutes (T3-12). After this time period, the study will be complete. A BIS value will be recorded before and after the dexmedetomidine bolus. The maintenance rate of TIVA will then be adjusted and further opioid given as per the anesthesiologist's preference, prior to and during surgery. NIBP readings will be recorded every 5 minutes throughout surgery and every 15 minutes in Post Anesthetic Care Unit (PACU), in addition to continuous ECG, HR and SpO2 monitoring.

Statistical Analysis The turning point estimator of Choi will be used to estimate the target dose. This describes how values of pairs at the crossover points are averaged. It is a form of target dose estimation that is frequently used in anesthesia UDM research.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Elective surgery
* Planned general anesthesia with TIVA
* Planned insertion of LMA
* Ages ≥ 5 to < 10 years

Exclusion Criteria:

* Cardiac disease
* Cardiac rhythm abnormalities
* Chronic hypertension
* Predicted difficult intubation
* Contraindication to LMA use
* Weight < 5th centile or > 95th centile for age
* Pre-operative administration of anxiolytics (such as benzodiazepines or opioid analgesics)
* Hypersensitivity to dexmedetomidine or any other study medication

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Dose of dexmedetomidine | 10 minutes for each patient
  Dose of dexmedetomidine that can be given as a rapid bolus that does not cause significant hemodynamic effects in healthy children

SECONDARY OUTCOMES:
BIS readings | 10 minutes for each patient
  Requirement for rescue intervention, BIS readings before and after dexmedetomidine bolus

CONTACTS AND LOCATIONS:
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada